CLINICAL TRIAL: NCT02838069
Title: A Phase IIb, Prospective, Multicentre, Double-blind, Triple-arm, Randomized Versus Placebo Trial, to Assess the Efficacy of a Single Injection of Either 2 or 10 x 106 Autologous Adipose Derived Mesenchymal Stromal Cells (ASC) in the Treatment of Mild to Moderate Osteoarthritis (OA) of the Knee, Active and Unresponsive to Conservative Therapy for at Least 12 Months
Brief Title: A Study Evaluating the Efficacy of a Single Injection Autologous Adipose Derived Mesenchymal Stromal Cells in Patients With Knee Osteoarthritis
Acronym: ADIPOA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Toulouse (Other); Assistance Publique - Hôpitaux de Paris (Other); National University of Ireland, Galway, Ireland (Other); Istituto Ortopedico Rizzoli (Other); Etablissement Français du Sang (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); European Clinical Research Infrastructure Network (Other); HUMAN MED AG (HM) (Unknown); Stichting Katholieke Universiteit (Other); SPORTS SURGERY CLINIC LIMITED (Unknown); University of Padova (Other); EVANGELISCHES WALDKRANKENHAUS SPANDAU KRANKENHAUSBETRIEBS GGMBH (EWK) (Unknown); PINTAIL LTD (PT) (Unknown); Centre National de la Recherche Scientifique, France (Other); University of Ulm (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Aries srl (ARIES) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL15_0453
Record Dates: First submitted 2016-06-13; First posted 2016-07-20 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2x106 ASC intra-articular injection (Experimental): Injection of Autologous adipose derived stem cells (2x106 ASC/5ml). The patient of this group will receive one single administration of the cells and will be followed for 12 months. A final follow up visit will occur at Month 24.
  Interventions: Biological: Injection (2x106 ASC/5ml).
- 10x106 ASC intra-articular injection (Experimental): Injection of Autologous adipose derived stem cells (10x106 ASC/5ml). The patient of this group will receive one single administration of the cells and will be followed for 12 months. A final follow up visit will occur at Month 24.
  Interventions: Biological: Injection (10x106 ASC/5ml).
- Placebo (Placebo Comparator): 0.5% glucose in saline with 4.5% albumin
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Injection (2x106 ASC/5ml). — Injection of Autologous adipose derived stem cells (2x106 ASC/5ml). The patient of this group will receive one single administration of the cells and will be followed for 12 months. A final follow up visit will occur at Month 24.
  Arms: 2x106 ASC intra-articular injection
Biological: Injection (10x106 ASC/5ml). — Injection of Autologous adipose derived stem cells (10x106 ASC/5ml). The patient of this group will receive one single administration of the cells and will be followed for 12 months. A final follow up visit will occur at Month 24.
  Arms: 10x106 ASC intra-articular injection
Other: Placebo — Injection of placebo 0.5% glucose in saline with 4.5% alb/5ml The patient of this group will receive one single administration and will be followed for 12 months. A final follow up visit will occur at Month 24.
  Arms: Placebo

SUMMARY:
ASCs will be administered via intra-articular use into the knee joint affected by OA where they are expected to exert their therapeutic effects.

The objective of this clinical trial is to generate efficacy and tolerability profiles of single injections of 2 dosages of autologous ASCs versus standard of care (placebo), when administered locally into a knee joint affected by OA after in vitro cell expansion. The potential of ASC to lead to a disease-modifying therapeutic option for the treatment of this chronic and debilitating disease will be assessed by MRI after 1 and 2 years.

This will be a phase IIb, multi-centre, prospective, randomized, double-blind study, comparing culture-expanded autologous ASC with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic mild to moderate osteoarthritis (OA) of the index knee as defined by the American college of Rheumatology (ACR)
* Must meet pain criteria at the time of screening/baseline visit since at least half of the days in the previous month
* NSAID washout of at least 2 days before screening/baseline

Exclusion Criteria:

* Previous treatments acting on cartilage or bone metabolism
* Received intra-articular injection of corticosteroids, platelet rich plasma or hyaluronic acid within the previous 6 months,
* Significant trauma or surgery to the index knee within the last year or arthroscopy of the index knee within 12 months of screening.
* Kellgren-Lawrence Grade 1 or 4 in the index knee on any incidences.
* Osteoarthritis causing significant pain in any joint other than the identified knee, i.e., pain in hip, or contralateral knee (≥ 20 mm pain) as confirmed by a separate VAS at baseline for any other painful joint concerned
* History of joint replacement of the knee or hip within the previous 12 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
Improvement of pain or physical function | Month 6
  evaluate the efficacy of ASC in mild to moderate knee OA (KL 2-3) based on increase in the number of "strict" responders defined by improvements from baseline in WOMAC pain or physical function subscores 50% with absolute changes 20 mm at 6 month, compared to placebo

SECONDARY OUTCOMES:
Disability (WOMAC) | Months 1, 3, 6, 12 and 24
  assessed by WOMAC questionnaire
Disability (KOOS) | Months 1, 3, 6, 12 and 24
  assessed by KOOS (Knee injury and Osteoarthritis Outcome Score questionnaire)
Disability (SAS) | Months 1, 3, 6, 12 and 24
  assessed by SAS questionnaire (The Short Arthritis Assessment Scale)
Change in Quality of life | Months 1, 3, 6, 12 and 24
  assessed by SF-36 questionnaire
painkillers consumption | Months 1, 3, 6, 12 and 24
  Changes from baseline (Day 0) to months 1, 3, 6, 12 and 24 in use of painkillers
Structural changes (X-Ray) | Months 12 and 24
  Changes from baseline (Day 0) to months 12 and 24 in femorotibial joint space of the index knee on X-ray
Structural changes (MRI) | Months 12 and 24
  Changes from baseline (Day 0) to months 12 and 24 by MOAKS (MRI Osteoarthritis Knee score)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jorgensen, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pers YM, Schrezenmeier H, Fleury-Cappellesso S, Noth U, Rackwitz L, Ferreira R, Berenbaum F, Ruyssen-Witrand A, Thurlings RM, Addimanda O, Lisignoli G, Ramonda R, Shannon F, Punzi L, Baillet A, McCaskie AW, McDonnell S, O'Callaghan J, Turmezei T, Kessler DA, Lotfi R, Rojewski M, Duffy A, Finnerty A, Moisan A, Brochot-Dechet H, Aubery-Rousselet M, Michon A, Bouzas-Rodriguez J, Pullig O, Broussous S, Nogue E, Amico M, Picot MC, Barry F, Jorgensen C; ADIPOA2 consortium. Effect of intra-articular adipose-derived mesenchymal stromal cell versus placebo injection on pain and function in patients with knee osteoarthritis: the ADIPOA2 phase 2b randomised clinical trial. Ann Rheum Dis. 2025 Dec;84(12):2103-2114. doi: 10.1016/j.ard.2025.07.026. Epub 2025 Aug 29. PMID 40885690